CLINICAL TRIAL: NCT02417194
Title: Prospective Cohort Study for the Impact of Preoperative Glycemic Control Status Measured by HbA1c Levels on Pathologic Features and Oncological Outcomes in the Patients With Renal Cell Carcinoma
Brief Title: Prognostic Significance of Preoperative Hemoglobin A1c (HbA1c) in Renal Cell Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Sung Kyu Hong, Associate professor, Seoul National University Bundang Hospital
Other Study IDs: L-2015-310
Record Dates: First submitted 2015-04-06; First posted 2015-04-15 (Estimated); Last update posted 2015-05-07 (Estimated); Status verified 2015-05

CONDITIONS: Carcinoma, Renal Cell; Pathology; Treatment Outcome; Hemoglobin A1c Protein, Human
Keywords: Renal cell carcinoma; hemoglobin A1c protein; Pathologic outcomes; Oncological outcomes; Nephrectomy
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
The effect of preoperative glycemic control measured by HbA1c on renal cell carcinoma (RCC) outcome remains controversial. Thus, the investigators aim to examine the association of preoperative glycemic control with oncologic outcomes after radical or partial nephrectomy. The investigators will prospectively collect the relevant data including preoperative HbA1c in 238 patients of RCC patients undergoing nephrectomy. The associations between clinical variables and risk of adverse pathological features and disease recurrence will be tested using a multivariate logistic regression and multiple Cox-proportional hazards model, respectively.

DETAILED DESCRIPTION:
* This is the observational study as the single institutional, prospective cohort study. The investigators prospectively collect the clinicopathological information of the patients with renal cell carcinoma (RCC) undergoing partial or radical nephrectomy.
* Particularly, the investigators check the variables, including age at surgery, body mass index, sex, comorbidities, preoperative HbA1c levels, blood urea nitrogen (BUN)/creatinine levels, estimated-GFR, clinical TMN staging by CT scan, final pathological results (TMN stage, histology, and Fuhrman nuclear grade), warm ischemic time and surgical margin status (in the case of partial nephrectomy), postoperative recurrence and distant metastasis, renal function changes during follow-up periods.
* The study protocol is same with routine follow-up schedule of the patients with RCC treated with nephrectomy. Typically, the investigators check the patients at 1, 3, 6, 12, 18, 24, 30 and 36 months. However, according to the patients status and preference, follow-up schedule can be changed within 3 months at specific time points. Because the present study is the observational cohort study, not intervention study, subtle changes of follow-up schedule would not affect on the primary outcomes.
* Importantly, preoperative HbA1c should be checked within 1 month before operation, same as the routine preoperative laboratory tests.

ELIGIBILITY:
Inclusion Criteria:

* Renal cell carcinoma (RCC) by image work-up such as CT scan
* Clinically localized RCC
* Aged over 20 years
* Patients undergoing radical or partial nephrectomy

Exclusion Criteria:

* distant metastasis, preoperatively
* preoperative targeted therapy
* preoperative immunotherapy
* medications affecting glucose status other than diabetes mellitus

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Enrolled patients should be diagnosed with renal cell carcinoma by ultrasonography and/or CT scan, MRI. In addition, the participants should be treated with radical or partial nephrectomy.
Sampling Method: Non-Probability Sample
Enrollment: 238 (Estimated)
Dates: Start 2015-04; Primary Completion 2018-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
TMN stage | within 2 weeks after surgery
  Pathological outcomes
Fuhrman (nuclear) grade | within 2 weeks after surgery
  Pathological outcomes
Recurrence-free survival | postoperative up to 3 years
  Oncological outcome: recurrence-free survival

SECONDARY OUTCOMES:
Postoperative renal function as assessed by estimated glomerular filtration rate (GFR) | postoperative up to 3 years
  estimated-GFR

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea